CLINICAL TRIAL: NCT05704478
Title: Impact of Vericiguat on Vascular Biology, as Well as Resting and Exertional Cardiovascular Performance Among Patients With Heart Failure With Reduced Ejection Fraction
Brief Title: Impact of Vericiguat on Hemodynamics of Heart Failure
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Basic Science
Other Study IDs: 22-2321
Record Dates: First submitted 2023-01-11; First posted 2023-01-30 (Actual); Last update posted 2025-11-13 (Actual); Status verified 2025-11

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure | interventions — vericiguat

STUDY DESIGN:
Intervention Model Description: Randomized clinical trial
Who Masked: Participant, Investigator
Masking Description: double-blind, both participant and provider. Blinding to be coordinated by research coordinator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (Active Comparator): Participants will be administered the drug vericiguat
  Interventions: Drug: Vericiguat
- Control (Placebo Comparator): Participants will be administered a placebo
  Interventions: Drug: Vericiguat

INTERVENTIONS:
Drug: Vericiguat — soluble guanylate cyclase stimulator

SUMMARY:
Vericiguat is a new drug that was recently approved by the Food and Drug Administration for patients with heart failure. In a large randomized controlled trial, this drug was found to help patients with heart failure live longer and stay out of the hospital more than normal treatment for heart failure. However, it is unclear how this drug positively impacts "hemodynamics", meaning how the heart functions during activity/exercise, and how it may also help blood pressure and health of the blood vessels and autonomic nervous system. This study, funded by the drug manufacturer, Merck Corp, will enroll 30 patients with heart failure. The patients will undergo baseline testing, and then be randomized to either receive vericiguat or a placebo for about three months, and then come back for follow-up testing to learn more about how the drug impacts heart function.

DETAILED DESCRIPTION:
Vericiguat is an oral soluble guanylate cyclase (sGC) stimulator, which enhances sGC sensitivity to nitric oxide (NO). Patients with heart failure with reduced ejection fraction (HFrEF) are known to have a reduction in NO bioavailability as a result of endothelial dysfunction, oxidative stress2 and presence of reactive oxygen species. In turn, there is a reduction in sGC activity, which is associated with multiple adverse cardiac effects, including cardiac stiffness and fibrosis, microvascular dysfunction and ultimately, propagation of HFrEF. In a large, multi-center randomized placebo controlled trial, vericiguat reduced the incidence of death from cardiovascular causes or hospitalization for heart failure. The VICTORIA trial demonstrated that on a larger scale (N=5050 patients), modulation of the NO-sGC pathway led to stabilization and improvement of the heart failure syndrome, which translated into improvements in hard outcomes.

There are a paucity of data, however, characterizing the direct effects of vericiguat on left ventricular function among humans suffering from HFrEF. The echocardiographic substudy of VICTORIA found that left ventricular ejection fraction (LVEF) improved from baseline to 8 months follow-up in both the placebo arm (31.8±8.2% to 34.2±9.2%, P<0.001) and the vericiguat arm (33.0±9.4% to 36.1±10.1%, P<0.001) and that LV end-systolic volume index (LVESVI) also declined in both arms. However, non-invasive, echocardiographic-derived metrics of ventricular function are relatively insensitive when compared to invasive determinants of overall cardiovascular performance. Thus, longitudinal changes in metrics such as LVEF and LVESVI, while informative, may not sufficiently characterize the physiologic adaptations that occur following modulation of the NO-sGC pathway, which in turn, translate into improvements in hard outcomes, which were observed in the VICTORIA trial.

The primary objective of this proposal is to precisely characterize the impact of NO-sGC modulation with the novel agent vericiguat on vascular biology, as well as resting and exertional cardiovascular performance among patients with heart failure with reduced ejection fraction (HFrEF). Our central hypothesis is that vericiguat improves endothelial function, which promotes arterial vasodilatation - and consequently, reduces left and right ventricular afterload. This reduction in afterload improves ventricular contractility, and in turn, reduces HFrEF severity by improving left and right-sided cardiovascular performance. This hypothesis will be tested through comprehensive assessment of longitudinal changes in vascular biology and cardiopulmonary performance among patients with HFrEF prior to, and following initiation of the novel oral sGC stimulator, vericiguat.

ELIGIBILITY:
Inclusion Criteria:

1. Adults 18 years of age or greater with New York Heart Association functional class II, III, or IV HFrEF with left ventricular ejection fraction < 45% within 12 months of enrollment;
2. elevated brain natriuretic peptide level (BNP) within 30 days of enrollment; and
3. history of worsening congestion, defined as a HF-hospitalization within 6 months of enrollment or increase in diuretic therapy without hospitalization within three months of enrollment.

Exclusion Criteria:

1. systolic blood pressure (SBP) below 100mmHg;
2. use of long-acting nitrates, soluble guanylate cyclase stimulators, or phosphodiesterase type 5 inhibitors;
3. use of intravenous inotropes or implantable left ventricular assist devices;
4. use of anticoagulants with an inability to temporarily hold these medications for procedures or to keep the international normalized ratio < 2.5 units;
5. uncontrolled arrhythmias;
6. noncardiac factors that may limit the ability to exercise (e.g. severe osteoarthritis, peripheral vascular disease, severe pulmonary disease); and
7. pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
cardiac output, L/min | 3 months
  cardiac output from heart catheterization

SECONDARY OUTCOMES:
Quality-of-life assessment | 3 months
  Kansas City Cardiomyopathy Questionnaire
oxygen uptake (VO2), ml/kg/min | 3 months
  Oxygen uptake during cardiopulmonary exercise testing
Pulmonary arterial pressure, mmHg | 3 months
  hemodynamics from heart catheterization
Pulmonary capillary wedge pressure, mmHg | 3 months
  hemodynamics from heart catheterization

CONTACTS AND LOCATIONS:
Locations (1):
- University of Colorado, Anschutz Medical Campus, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared with other researchers